CLINICAL TRIAL: NCT04941352
Title: The Effect of Interpersonal Relations Theory-Based Motivational Interviews on Functional Recovery and Insight Levels of Patients With Schizophrenia
Brief Title: Motivational Interviewing in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Nesrin Çunkuş, PhD student, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 60116787-020/50912
Record Dates: First submitted 2021-06-22; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Motivational Interviews; Schizophrenia
Keywords: Insight; Functional Recovery; Interpersonal Relations Theory; Motivational Interviews; Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Randomized controlled pre-post test design
Who Masked: Participant, Care Provider
Masking Description: Participants and caregivers were not informed about intervention content and measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Study group (Experimental): Study group intervention consists 6-session Interpersonal Relations Theory-Based Motivational Interviews and 3-month follow-up.
  Interventions: Behavioral: 6-session Interpersonal Relations Theory-based Motivational Interviews and 3 month follow-up.
- No Intervention: Control group (No Intervention): Control group receives general care and the training booklet at the end of the study. Also includes 3-month follow-up.

INTERVENTIONS:
Behavioral: 6-session Interpersonal Relations Theory-based Motivational Interviews and 3 month follow-up. — 6-session Interpersonal Relations Theory-based Motivational Interviews were applied to the individuals in the study group. All sessions were conducted face-to-face in the form of individual interviews. Each interview lasted an average of 30-40 minutes. With this intervention, it was aimed to increase treatment cooperation and motivation in individuals with schizophrenia, to increase insight, to improve adherence to treatment, daily living skills and social functionality.Study data were collected using a personal information form, the Functional Remission of General Schizophrenia Scale (FROGS) and the Scale for Assessing the Three Components of Insight (SAI). The data were analyzed on the basis of pre-intervention, post-intervention and 3 months after the intervention.
  Arms: Experimental: Study group

SUMMARY:
Introduction: A poor therapeutic relationship, low insight and lack of motivation are associated with poor adjustment (to symptoms, treatment, and environment) in patients with schizophrenia. In order to achieve better compliance and results, the therapeutic relationship and insight should be developed by increasing the motivation of individuals.

Purpose: This study examines the effect of Interpersonal Relations Theory-Based motivational interviews on functional recovery and insight levels of patients with schizophrenia.

Methods: This single-blind, randomized controlled study used the simple randomization method and employed a pretest-posttest control group design, which is an experimental research design. The study was conducted at Pamukkale University, Health Research and Application Center, Habib Kızıltaş Psychiatric Hospital from November 2019 to June 2020 and included 40 individuals (20 in the experimental and 20 in the control groups). Study data were collected using a personal information form, the Functional Remission of General Schizophrenia Scale (FROGS) and the Scale for Assessing the Three Components of Insight (SAI). The researchers carried out a 6-session Interpersonal Relations Theory-based motivational interview with the participants in the experimental group. No intervention was made to the control group. The data were analyzed on the basis of pre-intervention, post-intervention and 3 months after the intervention (follow-up).

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness that causes problems in the thoughts, feelings, and behaviors of the individual, impairs the ability to evaluate reality, has a unique world and keeps the individual away from social life, causes difficulties in his family and social environment, relapses, and is a progressive, severe mental illness when regular treatment is not applied.

It is reported that individuals diagnosed with schizophrenia have poor insight into how they evaluate the symptoms of the disease and what they expect from treatment. One of the problems of individuals diagnosed with schizophrenia is lack of motivation. It is stated that this may be caused by the dopaminergic system. This situation can cause individuals to have difficulties in social life.

In this context, it is important to evaluate motivational processes in the treatment of schizophrenia and to plan and implement initiatives that will increase motivation. A poor therapeutic relationship, low insight and lack of motivation are associated with poor adjustment (to symptoms, treatment, and environment) in patients with schizophrenia. In order to achieve better compliance and results, the therapeutic relationship and insight should be developed by increasing the motivation of individuals. Nurses need to establish a therapeutic relationship in order for the nursing care to produce effective results in the recovery process of these patients.

In this study, it is thought that Interpersonal Relations-Based Motivational Interviewing can be effective in increasing the symptom management, social-occupational functionality, adherence to treatment, daily life skills and insight levels of patients with schizophrenia, and may shed light and guide psychiatric nursing interventions.

ELIGIBILITY:
Inclusion Criteria:

* To be at least primary school graduate,
* Living in the city center of Denizli,
* Being open to communication and cooperation.
* Being between the ages of 18-65,
* Being in remission (period without psychotic exacerbation),
* To have a diagnosis of schizophrenia according to DSM-5 (The Diagnostic and Statistical Manual of Mental Disorders) diagnostic criteria.

Exclusion Criteria:

* Being under the age of 18 and over the age of 65,
* Being illiterate in Turkish,
* Having Mental Retardation,
* Being diagnosed with a mental illness other than schizophrenia according to the DSM-5 diagnostic criteria,
* Being in a psychotic attack period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Assessing the Three Components of Insight Score | Change from baseline Assessing the Three Components of Insight score at 3 months
  Scales were filled in by interviewing each participant. The scale consists of 8 questions. In the first 7 questions, each item is evaluated as 0-2. The highest total score of the first seven questions is 14. The eighth question is presented as an appendix. It is left to the researcher to ask this question. The highest total score with this question is 18. Increased score indicates an increase in insight.
Functional Remission of General Schizophrenia Score | Change from baseline Functional Remission of General Schizophrenia score at 3 months
  Scales were filled in by interviewing each participant. Scoring is done between 1-5 points. The maximum score that can be obtained from the scale is 95, and the minimum score is 19. Increased score indicates an increase in general functionality.

SECONDARY OUTCOMES:
Number of health care uses | Change in the number of initial health care use in the 3rd month
  According to the patient's declaration, number of hospitalizations.

CONTACTS AND LOCATIONS:
Overall Officials: Gülay Yiğitoğlu, PhD, Study Director — Pamukkale University; Nesrin Çunkuş, Msc, Principal Investigator — Pamukkale University; Ayşe Nur İnci Kenar, PhD, Study Chair — Pamukkale University
Locations (1):
- Pamukkale University Pamukkale University, Faculty of Health Science, Departmant of Psychiatric Nursing, Denizli, Kınıklı Kampus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study results will be announced in a publication.
Supporting Information: Study Protocol, SAP
Time Frame: Findings can be shared after the study has been published.
Access Criteria: The sociodemographic and disease-related characteristics of the participants, the pre-post-test and follow-up findings including the answers to the research questions and statistical analyzes will be shared.

REFERENCES:
- [Background] Townsend MC, Morgan KI. Schizoprenia spectrum and other Psychotic disorders. Psychiatric mental health nursing: Concepts of care in evidence-based practice. F. A. Davis Company, Philadelphia, 2017, s. 456-489.
- [Result] Medalia A, Brekke J. In search of a theoretical structure for understanding motivation in schizophrenia. Schizophr Bull. 2010 Sep;36(5):912-8. doi: 10.1093/schbul/sbq073. Epub 2010 Jun 30. PMID 20595203
- [Result] Pinho LGD, Pereira A, Chaves C. Nursing interventions in schizophrenia: The importance of therapeutic relationship. Nurse Care Open Acces J 2017; 3 (6): 331-333.
- [Result] World Health Organisation (WHO) 2019. Schizophrenia. [Last accessed on 2021 May 6]. Available from: https://www.who.int/news-room/fact-sheets/detail/schizophrenia
- [Result] Cho JM, Lee K. Effects of motivation interviewing using a group art therapy program on negative symptoms of schizophrenia. Arch Psychiatr Nurs. 2018 Dec;32(6):878-884. doi: 10.1016/j.apnu.2018.07.002. Epub 2018 Jul 19. PMID 30454632
- [Result] Fernandes MA, de Almeida JS, de Oliveira ÉKC, Sousa KHJF. Nursing process based on Peplau interpersonal relationship theory applied to schizophrenia. REUFPI 2018; 7 (3): 42-47.
- [Result] Ertem MY, Duman ZC. The effect of motivational interviews on treatment adherence and insight levels of patients with schizophrenia: A randomized controlled study. Perspect Psychiatr Care. 2019 Jan;55(1):75-86. doi: 10.1111/ppc.12301. Epub 2018 Jun 11. PMID 29888541